CLINICAL TRIAL: NCT06114719
Title: The Effect of Silymarin on the Prevention of Atrial Fibrillation After Coronary Artery Bypass Graft Surgery
Brief Title: Silymarin for the Prevention of Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Mihaela Preveden, Principal investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 661-1/1
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation New Onset
Keywords: cardiac surgery; postoperative atrial fibrillation; silymarin
MeSH Terms: interventions — Silymarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Silymarin 400 mg daily, orally, divided into two doses, for three days preoperatively
  Interventions: Drug: Silymarin
- Control group (No Intervention): Optimal standard therapy

INTERVENTIONS:
Drug: Silymarin — Subjects of the experimental group will receive silymarin (capsules containing 100 mg silymarin, expressed as silibinin) three days preoperatively. The dose they receive will be the recommended dose for the registered indications (400 mg daily, orally, divided into two doses).
  Arms: Experimental group

SUMMARY:
The study is a prospective, randomized, controlled trial to assess the effects of silymarin on the occurrence of postoperative atrial fibrillation after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a frequent complication after coronary artery bypass graft (CABG) surgery and is associated with increased mortality. So far, the effects of various drugs and supplements on the occurrence of postoperative atrial fibrillation (POAF) have been studied, but no one has looked into the effect of silymarin on the occurrence of POAF.

The study is designed as a prospective, randomized, controlled trial to assess the effects of silymarin on the occurrence of postoperative atrial fibrillation after CABG surgery. A total of 160 patients of both sexes scheduled for elective CABG surgery using cardiopulmonary bypass (CPB) will be included. They will be randomized into two groups (experimental and control) with 80 patients each. Subjects in the experimental group will receive 400 mg of silymarin three days preoperatively, while subjects in the control group will receive standard therapy.

The occurrence of POAF after CABG surgery will be the primary outcome, which will be defined as any dysrhythmia that represents the ECG characteristics of atrial fibrillation lasting at least 30 s on a rhythm strip or 12-lead ECG. Secondary outcomes will include postoperative values of inflammation markers, length of stay in the ICU, length of hospitalization, and occurrence of postoperative complications (pericardial effusion, stroke, in-hospital death).

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective CABG surgery using cardiopulmonary bypass
* first cardiac surgery
* left ventricular ejection fraction > 35%
* less than moderate mitral regurgitation

Exclusion Criteria:

* preoperative atrial fibrillation
* previous history of interventionally treated arrhythmias
* end-stage renal disease requiring hemodialysis
* chronic inflammatory and neoplastic diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative atrial fibrillation | 4 days
  Occurrence of postoperative atrial fibrillation lasting at least 30 s on a rhythm strip or 12-lead ECG

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Total duration of stay in the intensive care unit
Hospital length of stay | 30 days
  Total duration of stay in hospital
Postoperative complications | 30 days
  Occurrence of postoperative complications including pericardial effusion, stroke, and in-hospital death
Blood concentration of white blood cells | 4 days
  Postoperative values of white blood cells
Blood concentration of C-reactive protein | 4 days
  Postoperative values of C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Cardiovascular Diseases of Vojvodina, Kamenitz, Serbia